CLINICAL TRIAL: NCT01173692
Title: Minocycline for Reduction of Radiation Therapy Treatment-Related Symptom Burden in Oropharynx Cancer: A Randomized Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-0096; CA07 (Other: NCI); NCI-2012-01783 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Oropharynx Cancer
Keywords: Oropharynx Cancer; Radiation Therapy; XRT; Radiotherapy; Minocycline; Symptoms; Head and Neck
MeSH Terms: conditions — Oropharyngeal Neoplasms; cyclopia sequence | interventions — Minocycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Twice Daily Orally
  Interventions: Drug: Placebo
- Minocycline (Experimental): 100 mg Twice Daily Orally
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — 100 mg twice daily (200 mg) by mouth , every day for 7 weeks starting first day of radiation therapy.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Drug: Placebo — Twice daily by mouth, every day for 7 weeks starting at first day of radiation therapy.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if minocycline can reduce the symptoms reported by patients with oropharynx cancer, nasopharynx cancer, or unknown primary cancer of head and neck, who receive treatment with radiation therapy.

DETAILED DESCRIPTION:
The Study Drug:

Minocycline is an antibiotic and has been shown to interrupt cytokine production, which may help to reduce multiple symptoms.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Group 1 will take minocycline. Group 2 will take a placebo. A placebo is a substance that looks like the study drug but has no active ingredients.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take the study drug/placebo, by mouth, every day for 7 weeks starting at the first week of radiation therapy. You may take the study drug/placebo with a full glass (8 ounces) of water. You may take it with or without food. If it causes an upset stomach, you should take it with food. If you have trouble swallowing the dose of study drug/placebo, you can open the capsule right before you take them. You should not lie down for at least 30 minutes after taking the study drug/placebo to prevent possible irritation of the inside of the esophagus, a known side effect. You will be given pamphlets with more information about how to take the study drug/placebo.

You will be given a daily diary to write down what time you take the study drug/placebo. You must bring the diary with you to every study visit for the study doctor and research staff to review.

You must bring the study drug/placebo container to every study visit.

Study Visits:

Before you start your radiation treatment:

* You will have blood (about 2 teaspoons) drawn to check your liver function, if this test has not been done in the last 3 months.
* If you are able to become pregnant, you will have a urine pregnancy test. The study staff will give you the pregnancy test kit, and will review and record the results of the test before you can pick up the study drug from the pharmacy. If you are pregnant, you will not be given the study drug.
* You will also complete 5 questionnaires about pain and other symptoms, your alcohol and tobacco history, your health status, and your quality of life. It should take about 15 minutes to complete all of the questionnaires.

During radiation treatment (approximately Weeks 1- 7 of radiation):

You will complete the symptom questionnaire in the clinic or by telephone 2 times a week. You will be asked about symptoms you may be experiencing and how they may be interfering with your normal daily activities. You will complete the symptom questionnaire during one of your regular clinic visits. If you do not have a clinic visit scheduled around the time that the questionnaire needs to be completed, a member of the study staff will call you at your home at a time that is convenient for you. The symptom questionnaire should take about 5 minutes to complete each time.

At about Week 4 of radiation, you will complete 4 additional questionnaires about pain and other symptoms, your tobacco use, and a quality of life questionnaire. It should take about 5 minutes to complete all of the questionnaires.

During the last week of radiation (about Week 6-7), you will complete 4 additional questionnaires about pain and other symptoms, your health status, and your quality of life. It should take about 10 minutes to complete all of the questionnaires.

Starting after the last week of radiation (about Weeks 7-10), the study staff will call you 2 times each week to check on you. This phone call should last about 5 minutes. If you have had several side effects from the radiation therapy, this phone call may take longer.

Follow-Up Phone Calls:

During Weeks 11-15, you will complete the pain and other symptoms questionnaire 1 time a week by phone. A member of the study staff will call you at your home at a time that is convenient for you. The symptom questionnaire should take about 5 minutes to complete by phone each time.

End of Study Visit:

Your last study visit will be the same day that you have your last clinic visit with the radiation doctor (around Weeks 13-15). At this visit, you will complete the pain and other symptoms questionnaire, your health status and the 2 smoking questionnaires. It should take about 5 minutes to complete both questionnaires.

Length of Study:

You will be on study for up to 15 weeks. You will take the study drug/placebo for up to 7 weeks and continue to complete the symptom survey until 15 weeks. You will be taken off study early if you experience intolerable side effects or the study doctor thinks it is in your best interest.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Using minocycline for the treatment of the symptoms of radiation treatment for oropharynx cancer, nasopharynx cancer, or unknown primary cancer of head and neck, is investigational.

Up to 60 patients will take part in this research study. All will be enrolled at MD Anderson main campus as well as the regional care centers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of oropharyngeal cancer, nasopharyngeal cancer, or unknown primary cancer of head and neck in MDACC receiving radiation therapy with or without induction chemotherapy.
2. Patients > = 18 years old.
3. Patients with the above cancers, T0, TX, T1 to T3, N any, M0 receiving IMRT (to unilateral or bilateral neck) at least 64-72 Gy in 6-7 weeks as definitive treatment.
4. Patients must have normal renal function test and no prior renal disease: The screening cut off for serum creatinine < upper limit of normal.
5. Patients must have normal hepatic function test and no prior liver disease: The screening results for total bilirubin must be < 1.5 times the upper limit of normal. The screening results for the following must be < 2 times the upper limit of normal for patients to be eligible: Alkaline phosphatase (ALP) and Alanine aminotransferase (ALT). The screening results for Aspartate aminotransferase (AST) must be < 2 times the upper limit of normal if available.
6. Patients who speak English (due to the novel research and its complexity, we are only accruing English speaking patients to the protocol).
7. Patients must be willing to discontinue taking dong quai and/or St John's wort.
8. Patients must be willing and able to review, understand, and provide written consent.

Exclusion Criteria:

1. Patients receiving concurrent chemotherapy or concurrent biologic agent.
2. Patients who are taking medications or have conditions that potentially preclude use of any study medications or interventions as determined by the treating physician.
3. Patients who are enrolled in another symptom management trial or receiving active treatment under another clinical trial.
4. Bile duct obstruction or cholelithiasis.
5. History of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reaction.
6. Pre-existing psychosis or bipolar disorder.
7. Hypersensitivity to any tetracyclines.
8. Patients on anticoagulants (ie warfarin/heparin).
9. Patients with INR > 1.5.
10. Patients taking any tetracycline within the last 15 days.
11. Patients that are pregnant.
12. Patients treated with upfront radical surgery at the primary site (other than diagnostic tonsillectomy or excision).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07-22 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary B. Gunn, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 22, 2010 to Oct 10, 2013. All recruitment done at the University of Texas MD Anderson Cancer
Pre-assignment Details: 47 participants enrolled and assigned to the study drug. 7 participants withdraw after consent or within 2 weeks.
Groups:
- Minocycline: Minocycline 100mg (capsule) two times a day during the entire course of radiation therapy (7 weeks ± 5 days)
- Placebo: Placebo 100mg (capsule) two times a day during the entire course of radiation therapy (7 weeks ± 5 days)
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 22 | 25
Completed | 20 | 20
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Combined AUC for Selected Patient Symptoms
Description: 7-week (+/- 5 days) average area under the curve (AUC) for select MD Anderson Symptom Inventory for head and neck cancer (MDASI-HNC) symptoms namely fatigue, pain, sleep disturbance, difficulty swallowing and lack of appetite reported in the symptom survey. Each item is rated on a 11-point scale from 0 (not at all) to 10 (as bad as you can imagine). Higher values represent a worse outcome.
Time Frame: Up to 7 weeks
Population: Of 47 randomized patients, 40 (85% were evaluable for the primary efficacy analysis)
Measure: Mean (Standard Deviation); unit: score on a scale*week
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale*week | 3.1 (1) | 3.7 (1.7)

ADVERSE EVENTS:
Time Frame: From the start of the study medication, up to 30 days after last dose administered.
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=20) | Placebo (N=20)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT01173692/Prot_SAP_000.pdf